CLINICAL TRIAL: NCT06709287
Title: Comparison of Orthodontics Adverse Effects: Braces Versus Clear Aligners
Brief Title: Side Effects of Different Treatment Methods
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 17/2
Record Dates: First submitted 2024-10-15; First posted 2024-11-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Root Resorption; Pain; Chewing Function
Keywords: root resorption; pain; chewing function; fixed orthodontic treatment; clear aligner therapy
MeSH Terms: conditions — Root Resorption; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fixed orthodontic treatment: The patients in this group were treated with conventional braces.The patients were treated with 0.018-inch slot metal Roth brackets. Pretreatment (T0) digital lateral cephalometric radiographs were taken from the patients to compare pretreatment characteristics between the groups.The digital periapical radiographs taken with the paralleling technique were obtained.The digital periapical radiographs taken with the paralleling technique were obtained from the maxillary and mandibular incisors at the beginning of the treatment (T0) and after 6 months (T2).Probing depth, plaque index, and bleeding on probing were record at T0, after 3 months of treatment(T1), and at 6months(T2) to evaluate the periodontal status of the patients.A 5-question survey was used to evaluate pain levels, and a 9-question survey was used to evaluate chewing performance.
  Interventions: Other: orthodontic metal bracket
- clear aligners: The patients in this group were treated with clear aligners. Anterior teeth movement started from the first pair of aligners. Microfill and brace paste primers were used for bonding the attachments. Pretreatment (T0) digital lateral cephalometric radiographs were taken from the patients to compare pretreatment characteristics between the groups.The digital periapical radiographs taken with the paralleling technique were obtained.The digital periapical radiographs taken with the paralleling technique were obtained from the maxillary and mandibular incisors at the beginning of the treatment (T0) and after 6 months (T2).Probing depth, plaque index, and bleeding on probing were record at T0, after 3 months of treatment(T1), and at 6months(T2) to evaluate the periodontal status of the patients.A 5-question survey was used to evaluate pain levels, and a 9-question survey was used to evaluate chewing performance.
  Interventions: Other: clear aligners

INTERVENTIONS:
Other: clear aligners — The investigators measured pain and chewing performance at 8 time points during the first 6 months.
  Groups: clear aligners
Other: orthodontic metal bracket — Conventional metal bracket.
  Other Names: conventional bracket
  Groups: fixed orthodontic treatment

SUMMARY:
this study aimed to compare the effects of fixed orthodontic treatment and clear aligner therapy on root resorption, periodontal status, pain experience and chewing performance.

DETAILED DESCRIPTION:
The aim of the study is to compare the potential side effects of fixed orthodontic treatment and clear aligner therapy. 27 individuals who were treated with clear aligners (20 Female, 7 Male; mean age: 22.57 ± 7.37) and 22 patients treated with braces (14 Female, 8 Male; mean age: 17.05 ± 4.51) formed the study group. The periodontal statuses of the patients(Probing depth, bleeding on probing, plaque index) were evaluated before treatment (T0), 3 months (T1) after, and at 6th month (T2) following the beginning of the treatment. The amount of root resorption in maxillary & mandibular incisors was evaluated on periapical radiographies taken with the paralleling technique. Pain experience and chewing function were also recorded during treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with fixed braces or clear aligners
* patients with mild to moderate crowding
* patients without root canal treatment or resorption in anterior teeth
* patients with completed root development
* patients with good periodontal health at the beginning of the treatment
* patients with no congenitally missing or impacted tooth.

Exclusion Criteria:

* history of orthodontic therapy
* poor patient compliance
* presence of any craniofacial syndrome or systemic disease
* presence of cleft lip and palate
* trauma history
* mental retardation
* use of oral antiseptic solutions during orthodontic treatment
* need for scaling and root planning during treatment
* clear aligner patients with delayed movement of the anterior teeth.

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 22 patients (14 females, 8 males; mean age: 17.05 ± 4.51 years) who underwent fixed orthodontic therapy were included in the fixed treatment group and 27 patients (20 females, 7 males; mean age: 22.57 ± 7.37 years) who underwent clear aligner therapy were included in the clear aligner group.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
The primary outcomes of the study were pain scores and chewing performance scores. | 0-1 months
  The Visual Analog Scale has been used to evaluate pain scores and chewing performance. According to this scale, high scores represent good masticatory performance and high pain. Low scores represent poor masticatory performance and low pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided